CLINICAL TRIAL: NCT01494272
Title: Preemptive Analgesia in Children Using Caudal Epidural Ropivacaine: A Prospective, Randomized, Double-blinded, Controlled Study
Brief Title: Analgesia in Children Using Caudal Epidural Ropivacaine
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Shannon Mulder, MD, M.D., Loma Linda University
Other Study IDs: 5110235
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Inguinal Hernia; Circumcision
Keywords: caudal epidural analgesia; elective circumcision; elective inguinal herniorrhaphy
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group CB (Caudal Before-study group): This group will receive caudal ropivacaine and epinephrine after induction of general anesthesia prior to surgical incision
- Caudal After (CA)-control group: This group will receive caudal ropivacaine with epinephrine after completion of surgery but before emergence from anesthesia
- Local Infiltration After (LIA) control group: This group will receive local infiltration of ropivacaine around the surgery site at the conclusion of surgery but before emergence from anesthesia

SUMMARY:
Caudal epidural analgesia (caudal block)is used in standard pediatric anesthesia practice. It has been shown to be effective in managing postoperative pain in children undergoing abdominal and infraumbilical surgery (Tobias et al 1994). Furthermore, studies have shown that children receiving caudal blocks have secondary benefits such as lower narcotic and anesthetic requirements, more rapid awakening from general anesthesia, decreased time to discharge home, and fewer pain-related behaviors postoperatively (Conroy et al 1993, Tobias et al 1995, Tobias 1996).

This proposed study involves the use of a caudal block in children undergoing elective inguinal herniorrhaphy or orchiopexy to evaluate the role of preemptive analgesia in pediatric pain management. We hypothesize that by inhibiting peripheral pain receptors with a caudal block before the onset of a painful stimulus, we can decrease central nervous system sensitization and reduce postoperative analgesic requirements

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 months to 2 years
2. Weight 25kg or less
3. ASA class 1, 2, 3
4. Elective inguinal herniorrhaphy or orchiopexy

Exclusion Criteria:

1. Contraindications to caudal epidural analgesia
2. parent's refusal
3. skeletal or spinal cord anomaly
4. coagulopathy
5. infection at the insertion site
6. ongoing bacteremia
7. allergy to ropivacaine

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children under 2 years of age having an elective inguinal herniorrhaphy or orchiopexy.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Usage of pain medications | over 24 hours

SECONDARY OUTCOMES:
Pain scores | At various intervals for first 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Mulder, MD, Principal Investigator — Loma Linda University Medical Center
Locations (2):
- United States (2):
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University Outpatient Surgery Center, Loma Linda, California